CLINICAL TRIAL: NCT06768489
Title: A Phase 1b Study of JNJ-79635322 in Combination With Daratumumab With or Without Lenalidomide or in Combination With Pomalidomide for Multiple Myeloma
Brief Title: A Study of JNJ-79635322 in Combination With Daratumumab With or Without Lenalidomide or in Combination With Pomalidomide for Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 79635322MMY1002; 79635322MMY1002 (Other: Janssen Research & Development, LLC); 2024-515316-44-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment Regimen A and C: JNJ-79635322+Daratumumab (Experimental): Participants who have received 1-3 prior lines of therapy, including a proteasome inhibitor (PI) and an immunomodulatory drug (Treatment regimen A1) will receive a dose of JNJ-79635322 along with daratumumab to establish the recommended phase 2 doses (RP2D[s]) of the JNJ-79635322 during Part 1 (Dose Escalation) of the study. Based on the study evaluation team (SET) decision, enrollment may proceed in participants with newly diagnosed multiple myeloma (NDMM) (Treatment regimen A2/C). Dose escalation and de-escalation will be based on SET evaluation. In Part 2 (Dose Expansion) participants will receive a dose of JNJ-79635322 combination treatment regimen(s) at the RP2D(s) determined in Part 1 and in disease subgroup(s) to determine the safety and tolerability of the combination treatment regimens.
  Interventions: Drug: JNJ-79635322; Drug: Daratumumab
- Treatment Regimen B: JNJ-79635322+Pomalidomide (Experimental): Participants who have received greater than or equal to (>=)1 prior line of therapy, including a PI and lenalidomide, and are lenalidomide refractory or >=2 prior lines of therapy, including a PI and lenalidomide will receive a dose of JNJ-79635322 along with pomalidomide to establish the RP2D(s) of the JNJ-79635322 during Part 1 (Dose Escalation) of the study. Dose escalation and de-escalation will be based on SET evaluation. In Part 2 (Dose Expansion) participants will receive a dose of JNJ-79635322 combination treatment regimen(s) at the RP2D(s) determined in Part 1 and in disease subgroup(s) to determine the safety and tolerability of the combination treatment regimens.
  Interventions: Drug: JNJ-79635322; Drug: Pomalidomide
- Treatment Regimen D and E: JNJ-79635322 + Daratumumab + Lenalidomide Combination (Experimental): Participants with NDMM will receive a dose of JNJ-79635322 along with daratumumab and lenalidomide to establish the RP2D[s] of the JNJ-79635322 during Part 1 (Dose Escalation) of the study. Dose escalation and de-escalation will be based on SET evaluation. In Part 2 (Dose Expansion) participants will receive a dose of JNJ-79635322 combination treatment regimen(s) at the RP2D(s) determined in Part 1 and in disease subgroup(s) to determine the safety and tolerability of the combination treatment regimens.
  Interventions: Drug: JNJ-79635322; Drug: Daratumumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: JNJ-79635322 — JNJ-79635322 will be administered subcutaneously.
Drug: Daratumumab — Daratumumab will be administered subcutaneously.
  Arms: Treatment Regimen A and C: JNJ-79635322+Daratumumab; Treatment Regimen D and E: JNJ-79635322 + Daratumumab + Lenalidomide Combination
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Arms: Treatment Regimen B: JNJ-79635322+Pomalidomide
Drug: Lenalidomide — Lenalidomide will be administered orally.
  Arms: Treatment Regimen D and E: JNJ-79635322 + Daratumumab + Lenalidomide Combination

SUMMARY:
The primary purpose of this study for Part 1 (Dose Escalation) is to identify the safe effective dose (recommended Phase 2 doses [RP2Ds]) and schedule for JNJ-79635322 treatment regimen in combination with daratumumab with or without lenalidomide or with pomalidomide; and for Part 2 (Dose Expansion) is to further characterize the safety and tolerability of JNJ-79635322 combination treatment regimens at selected RP2D(s).

ELIGIBILITY:
Inclusion Criteria:

* Have documented initial diagnosis of multiple myeloma according to IMWG diagnostic criteria
* Meet treatment regimen-specific requirements as follows: Treatment regimen A (JNJ-79635322+daratumumab):Treatment regimen A1: Have been treated with 1 to 3 prior lines of therapy, including a proteasome inhibitor (PI) and an inhibitor, immunomodulatory drug (IMiD) therapy for the treatment of multiple myeloma (MM); Treatment regimen A2: Newly diagnosed MM naïve to multiple myeloma (or other related plasma cell neoplasm)-directed treatments; Treatment regimen B (JNJ-79635322+pomalidomide): Have received greater than or equal to (>=) 1 prior line of therapy, including a PI and lenalidomide, and are lenalidomide refractory OR >=2 prior lines of therapy, including a PI and lenalidomide; Treatment Regimens C, D, and E: Newly diagnosed MM naïve to multiple myeloma (or other related plasma cell neoplasm)-directed treatments
* Have a weight >=40 kilograms
* Must have an Eastern Cooperative Oncology Group status of 0 or 2
* Have measurable disease at screening as defined by at least 1 of the following: a) Serum monoclonal protein (M-protein) level >= 0.5 gram per deciliter (g/dL); or b) Urine M-protein level >=200 milligram (mg)/24 hours; or c) Light chain multiple myeloma: Serum immunoglobulin (Ig) free light chain (FLC) >= 10 mg/dL and abnormal serum Ig kappa lambda FLC ratio. d) For participants without measurable disease in the serum, urine, or involved FLC: presence of 1 or more focus of extramedullary disease which meets the following criteria: extramedullary plasmacytoma not contiguous with a bone lesion, at least 1 lesion >=2 centimeter (cm) (at its greatest dimension) diameter on whole body positron emission tomography-computed tomography (or whole-body magnetic resonance imaging approved by sponsor), and not previously radiated

Exclusion Criteria:

* Any serious underlying medical conditions, such as: a) Evidence of active viral, bacterial, or systemic fungal infection requiring ongoing antiviral, antibacterial, or antifungal treatment. b) Active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before start of study treatment. c) Cardiac conditions (myocardial infarction, unstable angina, or coronary artery bypass graft <=6 months prior to enrollment; New york heart association stage III or IV congestive heart failure et cetera)
* Prior antitumor therapy as follows, in the specified time frame prior to the first dose of study treatment: a) Targeted therapy, epigenetic therapy, monoclonal antibody (mAb) treatment, or treatment with an investigational drug or an invasive investigational medical device within 21 days or 5 half-lives, whichever is less. b) Gene-modified adoptive cell therapy (example, chimeric antigen receptor [CAR] modified T cells, natural killer cells) within 90 days. c) Prior anti-CD38 directed therapy within 90 days (for treatment regimen A only; within 21 days for treatment regimen B). d) Conventional chemotherapy within 21 days. e) PI therapy within 14 days. f) Immunomodulatory agent therapy within 7 days. g) Radiotherapy within 14 days
* Stem cell transplantation: a) Allogeneic stem cell transplant within 6 months before the first dose of study treatment. b) Received an autologous stem cell transplant less than or equal to (<=)12 weeks before the first dose of study treatment
* Nonhematologic toxicity from prior anticancer therapy that has not resolved to baseline level or to grade <=1 (except alopecia, tissue post-RT fibrosis [any grade] or peripheral neuropathy grade <=3)
* Prior treatment with CD3-redirecting therapy
* The following medical conditions: pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation, human immunodeficiency (HIV) infection, active hepatitis B or C infection, stroke or seizure within 6 months prior to first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 28 days
  DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Number of Participants with Adverse Events (AEs) by Severity | Up to 3 Years and 3 months
  An AE is any untoward medical occurrence in a clinical study participant that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.
Number of Participants with Clinically Significant Laboratory Abnormalities | Up to 3 Years and 3 months
  Participants with clinically significant laboratory abnormalities (hematology and chemistry) will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response Rate | Up to 3 Years and 3 months
  Overall response rate is defined as percentage of participants who have a partial response (PR) or better evaluated by the investigator as per international myeloma working group (IMWG) 2016 criteria.
Duration of Response (DOR) | Up to 3 Years and 3 months
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), as per IMWG 2016 response criteria, or death due to progression, whichever occurs first.
Time to Response (TTR) | Up to 3 Years and 3 months
  TTR is defined as the time between date of first dose of study treatment and the first efficacy evaluation at which the participant has met all criteria for PR or better as defined by IMWG 2016 response criteria.
Serum Concentration of JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  Serum samples will be analyzed to determine concentrations of JNJ-79635322 and daratumumab.
Area Under the Serum Concentration Time Curve from Time Zero to Infinity (AUCinf) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  AUCinf for JNJ-79635322 and daratumumab will be reported.
Area Under the Serum Concentration Time Curve from Time Zero to the Last Measurable Concentration [AUC(0-t)] for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  AUC(0-t) for JNJ-79635322 and daratumumab will be reported.
Area Under the Serum Concentration Time Curve During the Dosing Interval (AUCtau) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  AUCtau for JNJ-79635322 and daratumumab will be reported.
Maximum Serum Concentration (Cmax) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  Cmax for JNJ-79635322 and daratumumab will be reported.
Half Life (T1/2) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  T1/2 for JNJ-79635322 and daratumumab will be reported.
Time to Reach Cmax (Tmax) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  Tmax for JNJ-79635322 and daratumumab will be reported.
Systemic Clearance (CL/F) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  CL/F for JNJ-79635322 and daratumumab will be reported.
Apparent Volume of Distribution at Steady State (Vss/F) for JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  Vss/F for JNJ-79635322 and daratumumab will be reported.
Number of Participants with Presence of Anti-Drug Antibodies to JNJ-79635322 and Daratumumab | Up to 3 Years and 3 months
  Participants with anti-drug antibodies to JNJ-79635322 and daratumumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- Australia (5):
  - Monash Medical Centre, Clayton
  - St Vincents Hospital Melbourne, Fitzroy
  - Peter MacCallum Cancer Centre, Melbourne
  - Calvary Mater Newcastle Hospital, Waratah
  - Wollongong Hospital, Wollongong
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Spain (2):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Pillarisetti K, Yang D, Luistro L, Yao J, Smith M, Vulfson P, Testa J Jr, Ponticiello R, Brodeur SR, Heidrich B, Packman K, Singh S, Attar RM, Elsayed YA, Philippar U. Ramantamig (JNJ-79635322), a novel T-cell-engaging trispecific antibody targeting BCMA, GPRC5D, and CD3, in multiple myeloma models. Blood. 2025 Oct 16:blood.2025030027. doi: 10.1182/blood.2025030027. Online ahead of print. PMID 41100731